CLINICAL TRIAL: NCT03194581
Title: Normoxic Challenges Utility to Evaluate Blood Loss Through Cerebral Oxygenation
Brief Title: Normoxic Challenges Utility to Evaluate Blood Loss
Status: Terminated | Type: Observational
Why Stopped: Profissional reasons, not related with the study
Sponsor: Centro Hospitalar do Tâmega e Sousa (Other)
Responsible Party: Principal Investigator, Mariana Marques da Cunha, MD, Centro Hospitalar do Tâmega e Sousa
Other Study IDs: HEMOX
Record Dates: First submitted 2017-06-12; First posted 2017-06-21 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cerebral oxygenation — Evaluate cerebral oxygenation using normoxic challenges

SUMMARY:
This study will evaluate the impact of repeated normoxic challenges on cerebral oxygenation as a measure of the effect of blood loss on DO2 during surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* High risk of intraoperative blood loss
* General anaesthesia

Exclusion Criteria:

* Respiratory insufficiency
* Ischemic heart disease
* Stroke
* ASA classification > 3
* Laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to surgery with high risk of blood loss
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in cerebral regional oxygen saturation | Before and 3 minutes after normoxic challenges

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Tâmega e Sousa, Penafiel, Porto District, Portugal